CLINICAL TRIAL: NCT04756076
Title: Study Roles of Heavy Metals and Essential Metal Dyshomeostasis in Pulmonary Arterial Hypertension Patients
Status: Recruiting | Type: Observational
Sponsor: Jiapeng Huang (Other)
Responsible Party: Sponsor-Investigator, Jiapeng Huang, Principal Investigator, University of Louisville
Organization: University of Louisville (Other)
Other Study IDs: 20.0947
Record Dates: First submitted 2021-02-07; First posted 2021-02-16 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Hypertension; Metal Poison
MeSH Terms: conditions — Hypertension, Pulmonary; Heavy Metal Poisoning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: age and gender matched controls
  Interventions: Diagnostic Test: Metal level measurements
- Pulmonary Hypertension Group: Pulmonary Hypertension Patients with Various Degree of Severity
  Interventions: Diagnostic Test: Metal level measurements

INTERVENTIONS:
Diagnostic Test: Metal level measurements — Measure multiple metal levels

SUMMARY:
Investigators plan to recruit 50 PAH patients from UofL PAH Clinic, with various degrees of severity (25 intermediate risk patients and 20 high risk patients) and 10 age and gender matched controls. PAH patients are evaluated at least every 6 months by the PAH Clinic and blood/urine samples will be obtained at each office visit. Blood, plasma and urine samples will be used to measure 31 metal levels including heavy metals (cadmium, arsenic, cobalt, lead etc.) and essential metals (calcium, copper, iron, zinc, potassium etc.) by the with ICP-MS via the service of ITEMFC. Interactions among the 31 metals in PAH patients, metal concentration differences between intermediate risk PAH, high risk PAH and control groups, the correlation between metal concentrations and the etiology, severity, duration, treatment, and progression of PAH/RV dysfunction over 12 months will be analyzed by CIEHS Biostatistics and Informatics Facility Core.

DETAILED DESCRIPTION:
Exposures to heavy metals such arsenic, lead, cadmium have been linked to increased incidence of cardiovascular disease (CVD). However, current studies suffer from multiple drawbacks, most studies were cross sectional in design, focused on individual metals without consideration of the joint effects of multiple metals, and did not examine the possible effects of essential metals in CVD. Especially, the relationship between heavy metals/essential metal dyshomeostasis and right ventricular (RV) dysfunction/pulmonary hypertension (PAH), is less investigated. Investigators hypothesize that increased toxic heavy metals and/or essential metal dyshomeostasis impact hypoxia response, endothelial dysfunction, perivascular inflammation and vascular remodeling of the pulmonary vasculature, and are important pathogenic initiators/stimulators during the progression of PAH and associated RV remodeling/dysfunction.

Investigators plan to recruit 50 PAH patients from UofL PAH Clinic, with various degrees of severity (25 intermediate risk patients and 20 high risk patients) and 10 age and gender matched controls. PAH patients are evaluated at least every 6 months by the PAH Clinic and blood/urine samples will be obtained at each office visit. Blood, plasma and urine samples will be used to measure 31 metal levels including heavy metals (cadmium, arsenic, cobalt, lead etc.) and essential metals (calcium, copper, iron, zinc, potassium etc.) by the with ICP-MS via the service of ITEMFC. Interactions among the 31 metals in PAH patients, metal concentration differences between intermediate risk PAH, high risk PAH and control groups, the correlation between metal concentrations and the etiology, severity, duration, treatment, and progression of PAH/RV dysfunction over 12 months will be analyzed by CIEHS Biostatistics and Informatics Facility Core.

Heavy metals have the potential of generating reactive oxygen species (ROS) and oxidative stress whenever the release of ROS exceeds endogenous antioxidant capacity. Therefore, investigators hypothesize that heavy metal/essential metal dyshomeostasis could induce oxidative stress responses, activate two key pulmonary vasculature regulators (endothelin 1 and hypoxia inducible factor (HIF) pathways), and in turn contributes to the PAH pathogenesis and RV dysfunction. Oxidative stress, endothelin 1 and HIF pathway markers in the blood will be measured with ELISA kits in both PAH and control groups. Investigators will perform comprehensive correlation analysis between metal levels, oxidative stress markers, endothelin 1 and HIF pathway markers, and quantitative clinical biomarkers such as hemodynamic, laboratory and functional data in PAH patients. Furthermore, investigators will perform correlation analysis between blood levels of oxidative stress, endothelin 1 and HIF pathway markers and the patients' dietary intake of antioxidant vegetables.

ELIGIBILITY:
Inclusion Criteria:

* All patients with the diagnosis of pulmonary hypertension
* Agree to the study protocol
* Healthy volunteers
* Age, gender matched controls

Exclusion Criteria:

* Younger than 18 years
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Metal levels in control and pulmonary hypertension groups | up to 12 months
  Metal levels in control and pulmonary hypertension groups

SECONDARY OUTCOMES:
Right heart catheterization data | up to 12 months
  mean pulmonary artery pressure (mmHg)
Pulmonary hypertension risk scores (Registry to Evaluate Early and Long-Term PAH Disease Management) | up to 12 months
  Pulmonary hypertension risk scores, 0-10, the higher score means a worse outcome.
Mortality | up to 12 months
  death

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville Health, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No